CLINICAL TRIAL: NCT02140424
Title: Bone Mineral Accrual and Microarchitecture in Youth With Type 1 Diabetes
Brief Title: Bone Health in Youth With Type 1 Diabetes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Deborah Mitchell, MD, Assistant Professor in Pediatrics, Massachusetts General Hospital
Other Study IDs: 2013P000985
Record Dates: First submitted 2014-05-13; First posted 2014-05-16 (Estimated); Last update posted 2020-10-09 (Actual); Status verified 2020-10

CONDITIONS: Type 1 Diabetes; Osteoporosis
Keywords: type 1 diabetes; osteoporosis; children
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Osteoporosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum, plasma, urine
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- youth with type 1 diabetes
- healthy controls

SUMMARY:
This is an observational study of children and young adults ages 6-20 years with type 1 diabetes and age- and race-matched controls. The investigators will be examining blood and urine hormone levels as well as measures of bone density including DXA and high-resolution peripheral quantitiative computed tomography. The investigators will also be collecting data regarding physical activity via use of wearable accelerometers. The investigators hypothesize that youth with type 1 diabetes will have slower bone accrual and impaired bone microarchitectural integrity compared with non-diabetic controls, and that bones of individuals with type 1 diabetes will not respond as well to physical activity. The investigators hypothesize that poor bone accrual will be associated with sub-optimal glucose control as well as lower levels of insulin-like growth factor 1.

ELIGIBILITY:
Inclusion Criteria:

* Age 6-20 years
* Out of honeymoon period (cohort with diabetes)

Exclusion Criteria:

* BMI<5th percentile for age
* BMI>95th percentile for age
* Celiac disease
* Hyperthyroidism, uncontrolled hypothyroidism
* History of significant hepatic disease, renal disease, oncologic disease, cardiovascular disease, psychiatric disease
* Anemia (Hgb <11)
* Taking medications other than insulin known to affect bone health (including hormonal contraception, glucocorticoids, growth hormone)

Ages: 6 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: youth and young adults with type 1 diabetes and healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 242 (Estimated)
Dates: Start 2013-08; Primary Completion 2023-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Rate of bone mineral accrual | 0, 12, 24 months
  Bone mineral mass and density will be measured by dual-energy x-ray absorptiometry (DXA) at baseline and 12 months. Percent change over time will be calculated and then compared in subjects with type 1 diabetes and matched control subjects.

SECONDARY OUTCOMES:
Cross-sectional comparison of bone microarchitectural parameters in patients with diabetes vs. controls | Baseline
  Bone microarchitecture will be assessed by high-resolution peripheral quantitative computed tomography (HR-pQCT). Parameters measured will include cortical compartment density, cortical thickness, cortical porosity, trabecular density, trabecular number, and trabecular thickness.
Rate of bone mineral accrual | 0 and 24 months
  Bone mineral mass and density will be measured by dual-energy x-ray absorptiometry (DXA) at baseline and 24 months. Percent change over time will be calculated and then compared in subjects with type 1 diabetes and matched control subjects.
Change bone microarchitectural parameters in patients with diabetes vs. controls | 0 and 24 months
  Bone microarchitecture will be assessed by high-resolution peripheral quantitative computed tomography (HR-pQCT) at 0 and 12 months. Parameters measured will include cortical compartment density, cortical thickness, cortical porosity, trabecular density, trabecular number, and trabecular thickness and percent change over 12 months will be calculated. Percent change will be compared in patients with diabetes and matched controls.

OTHER OUTCOMES:
Association of glycemic control with bone mineral accrual | 0 and 24 months
  Glycemic control will be assessed by hemoglobin A1c measurements at study visits and as part of routine diabetes care. An average hemoglobin A1c over the time of observation will be calculated using the trapezoidal rule. Association of glycemic control with bone mineral accrual as measured by DXA will be examined via regression analysis.
Association of bone mineral accrual with moderate-to-vigorous physical activity | 0 and 24 months
  activity will be assessed with accelerometers. The association of bone accrual among youth with and without diabetes will be assessed by correlation analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Deborah M Mitchell, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Joseph TV, Caksa S, Misra M, Mitchell DM. Hip Structural Analysis Reveals Impaired Hip Geometry in Girls With Type 1 Diabetes. J Clin Endocrinol Metab. 2020 Dec 1;105(12):e4848-56. doi: 10.1210/clinem/dgaa647. PMID 32929477
- [Derived] Mitchell DM, Caksa S, Joseph T, Bouxsein ML, Misra M. Elevated HbA1c Is Associated with Altered Cortical and Trabecular Microarchitecture in Girls with Type 1 Diabetes. J Clin Endocrinol Metab. 2020 Apr 1;105(4):e1648-56. doi: 10.1210/clinem/dgz221. PMID 31761940